CLINICAL TRIAL: NCT00708786
Title: Ventricular Arrhythmias Incidence According to Sleep Apnea Syndrome in ICD Patients
Brief Title: Ventricular Arrhythmias Incidence According to Sleep Apnea Syndrome in Implantable Cardioverter-Defibrillator (ICD) Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LivaNova (Industry)
Responsible Party: F. Anselme - Principal investigator, CHRU Charles Nicolle
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITAC01-VISION
Record Dates: First submitted 2008-04-07; First posted 2008-07-02 (Estimated); Last update posted 2008-07-02 (Estimated); Status verified 2008-06

CONDITIONS: Sleep Apnoea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: ICD — Ventricular arrhythmia treatment
Device: CRT-D — Ventricular arrhythmia treatment

SUMMARY:
The purpose of this study is to report the incidence of ventricular arrhythmias correlated to the SAS and to focus on the interest of diagnosing Sleep-disorders breathing in ICD patients. This diagnosis will be assessed by an ambulatory nasal pressure recording with portable multi-channel recorder associated to a complete SAS related symptoms questionnaire.This clinical trial will be the first step to gather information about the suspected sleep relation between ventricular arrhythmias and Sleep breathing disorders, in order to improve the management and treatment of such arrhythmias in next generation of defibrillators which will integrate a minute ventilation sensor able to monitor breathing.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are at risk of sudden death due to ventricular arrhythmia and who satisfy at least one of the following criteria are eligible for enrolment:
* Class I indications for ICD

  * Survival of at least one episode of cardiac arrest due to VT or VF not due to a transient or reversible cause, or presumed to be due to VF when electrophysiological testing is precluded by other medical conditions; or
  * Spontaneous sustained ventricular tachycardia, or
  * Syncope of undetermined origin with clinically relevant haemodynamically significant sustained VT or VF induced at electrophysiological study when drug therapy is ineffective, not tolerated or not preferred, or
* Class IIa Indication for ICD

  * Non-sustained VT with coronary disease, prior myocardial infarction, left ventricular dysfunction (≤ 40%) and inducible VF or sustained VT at electrophysiological study.
  * With prior myocardial infarction and LVEF less than 30 % (without prior life-threatening arrhythmia or sustained VT).
* Patients candidate for cardiac resynchronization therapy (CRT) need to be in functional Class III or IV of the NYHA classification.

Patients will be included only after having granted their informed consent to participate in the study, preceded by the delivery of appropriate information

Exclusion Criteria:

* VT/VF is associated with drug toxicity, electrolyte imbalance, hypoxia, electrocution or other reversible cause;
* VT/VF occurred during the acute phase of infarction (< 1 week) or during an unstable ischemic phase;
* Incessant VT/VF;
* Implanted pacemaker that is not going to be explanted or otherwise disabled;
* Inability or refusal to provided informed consent
* Tricuspid valvular disease or tricuspid mechanical heart valve (lead contraindication);
* Unable to understand the purpose and plan of the study;
* Geographically unstable or not available for follow-up as defined in the investigational plan;
* Reduced life expectancy (≤ 1 year) for other than cardiovascular reasons;
* Patient participating in another clinical study;
* Patient of minor age (< 18 years);
* Pregnancy (Women of childbearing potential are required to have a negative pregnancy test within seven days prior to enrollment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 755 (Estimated)
Dates: Start 2004-04; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to assess the correlation between ventricular arrhythmias and Sleep apnoea syndrome in ICD patients during a 12-month follow-up. | 12 months

SECONDARY OUTCOMES:
To determine the number of arrhythmias in the morning (between 06:00 and 12:00 AM). The circadian distribution of global arrhythmias will be presented. | 12 months
To report and compare the number of hospitalizations, mortality, and morbidity according to Respiratory Disturbance Index (RDI). | 12 months
To evaluate the incidence of adverse events in the studied population: device-related adverse events with an actual or potential effect on the patient, serious adverse events not related to the device, mortality, and unanticipated adverse device effects | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Anselme, MD, Principal Investigator — CHU Charles Nicolle - Rouen
Locations (30):
- France (19):
  - CHRU Hopital de la cavale blanche, Brest
  - CHU, Clermont-Ferrand
  - CHU - Hopital Michallon, Grenoble
  - CHU Dupuytren, Limoges
  - Hopital cardiologique, Lyon
  - Hopital Saint Joseph et saint Luc, Lyon
  - Hopital Nord, Marseille
  - CHR Notre Dame de Bonsecours, Metz
  - CH Montpellier, Montpellier
  - Nouvelle Clinique Nantaise, Nantes
  - Clinique Bizet, Paris
  - CH Pau, Pau
  - CHU Hopital la Milétrie, Poitiers
  - CHR Cardiologie A, Rennes
  - CHU Charles Nicolle, Rouen
  - Clinique Pasteur, Toulouse
  - CHRU Hopital Trousseau, Tours
  - Clinique Saint gatien, Tours
  - CHRU Brabois, Vandœuvre-lès-Nancy
- Germany (3):
  - Herz-Kreislauf-Klinik Bevensen AG, Bad Bevensen
  - Universitatsklinikum Hamburg Eppendorf, Hamburg
  - Prof. Frey Praxis Starnberg, Starnberg
- Onassis Cardiac Surgery Center, Athens, Greece
- Italy (7):
  - Ospedale Mellini, Chiari (BS)
  - Osp. Civile, Desio
  - Casa di Cura Montevergine, Mercogliano
  - Policlinico de Modenna, Modenna
  - Instituto di Cura, Pavia
  - Hospitale civile Guglielmo da Saliceto, Piacenza
  - Policlinico San Donato, San Donato